CLINICAL TRIAL: NCT03213847
Title: Superb Microvascular Imaging of Median Nerve in Carpal Tunnel Syndrome: A Novel Technique in Diagnostic Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Ali Yavuz Karahan, Associate professor, Uşak University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMI001
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Carpal Tunnel Syndrome Bilateral
Keywords: Carpal Tunnel Syndrome; Superb microvascular imaging; Doppler ultrasound; Ultrasound; Median Nerve Entrapment; Diagnoses Disease
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with carpal tunnel syndrome (Other): Participants diagnosed with carpal tunnel syndrome; will be evaluated with Doppler ultrasound and superb microvascular imaging (SMI) ultrasound. The results of these two evaluations will be compared between each other in according to severity of carpal tunnel syndrome (severity will be determined by electromyography studies)
  Interventions: Device: Superb microvascular imaging (SMI) (Toshiba)

INTERVENTIONS:
Device: Superb microvascular imaging (SMI) (Toshiba) — to determine whether there is a correlation between the increased intraneural flow as measured using Doppler US and SMI methods and the severity of CTS as measured by nerve conduction studies, we designed this study

SUMMARY:
The aim of the study was to determine whether there is a correlation between the increased intraneural flow as measured using Doppler ultrasound (US) and superb microvascular imaging (SMI) methods and the severity of CTS as measured by nerve conduction studies. Moreover, investigators investigated the association of increased intraneural flow with the cross sectional area of the median nerve. The null hypothesis that there is no correlation between increased intraneural flow and the severity of carpal tunnel syndrome.

DETAILED DESCRIPTION:
Thanks to ultrasound (US) has a low cost, portable, available and non-invasive, the use of diagnostic US in musculoskeletal diseases is rapidly growing in worldwide. Because it is easy to identify the limb structures such as muscle, tendon, and nerves and also, their pathologies, US is frequently used by physiatrists, orthopedics, rheumatologists, sports medicine and pain management physicians nowadays. Providing images of the median nerve (MN) and accompanying structures and give dynamic images about the anatomy of the carpal tunnel are the most superiorities of US in carpal tunnel syndrome (CTS) diagnosis. The diagnose of CTS based on history and physical examination and confirmed with electrodiagnostic studies. Although the specificity of nerve conduction tests is high, there is significant variability in sensitivity (62-85%). Therefore, US has been suggested as an additional or alternative diagnose of CTS. Especially measurement of the cross-sectional area (CSA) of the MN is significantly greater in CTS patients and shows a significant correlation with electrodiagnostic findings such as sensory nerve conduction velocity (SCV) and distal motor latency (DML). Because it enhances the diagnostic accuracy the detection of the epineural or intraneuronal blood flow, the three techniques of Doppler US, are more recently preferred. The contributions of color, power and spectral Doppler techniques in CTS diagnosis, were studied in various studies before. While for the detection of intraneural flow, the power Doppler (PD) seems to be the best way, the specify, sensitivity and diagnostic accuracy of each Doppler techniques were good in most studies.

Superb microvascular imaging (SMI) (Toshiba Medical Systems, Tokyo, Japan) is a new era in diagnostic ultrasound image processing technique. This new technology assigns accurate visualization of vascular structures with intensive clutter suppression to provide flow signals large to small vessels and represent this data at high frame rates. The both of the two modes (color SMI (cSMI) and the monochrome SMI (mSMI)) of the SMI, allows to visualizing lower velocity blood flows and smaller vessels without the use of contrast medium. To the best of our knowledge, there have been no clinical trials which studied of the healthy or injured median nerve blood flow with SMI.

The aim of the study was to compare the diagnostic value of Doppler US and SMI methods in CTS based on detection of increased intraneural flow. Moreover, investigators investigated the association of increased intraneural flow with the CSA of the MN. The null hypothesis that there is no difference between Doppler US and SMI methods in the detection of increased intraneural flow in CTS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed as as mild, moderate or severe CTS with electromyography
* Age between 18-45

Exclusion Criteria:

* History of upper extremity trauma
* Diabetes mellitus
* Pregnancy,
* Rheumatological diseases
* Hypothyroidism

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-25 (Actual)

PRIMARY OUTCOMES:
Vascular blood flow images from median nerve (enterrapted in carpal tunnel) obtained with Power Doppler and Superb microvascular imaging. | Each participant will be assessed only one time at the admission time to the outpatient clinic
  Four-stage classify will be use for grading these images; Grade 0: No vascularity in MN, Grade 1: One or two focal color-encoded spots in MN, Grade 2: One linear color-encoded line or more than two focal color-encoded spots in MN, Grade 3: More than one linear color-encoded line in MN

CONTACTS AND LOCATIONS:
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Anthropometric and demographic data included age, weight, height, body mass index (BMI), gender, occupation, medication history and hand dominance. Main outcomes of the study: correlation between the increased intraneural flow as measured using Doppler US and Superb microvascular imaging (SMI) methods.

REFERENCES:
- [Background] Orlandi D, Gitto S, Perugin Bernardi S, Corazza A, De Flaviis L, Silvestri E, Cimmino MA, Sconfienza LM. Advanced Power Doppler Technique Increases Synovial Vascularity Detection in Patients with Rheumatoid Arthritis. Ultrasound Med Biol. 2017 Sep;43(9):1880-1887. doi: 10.1016/j.ultrasmedbio.2017.05.004. Epub 2017 Jun 17. PMID 28629689
- [Background] Akcar N, Ozkan S, Mehmetoglu O, Calisir C, Adapinar B. Value of power Doppler and gray-scale US in the diagnosis of carpal tunnel syndrome: contribution of cross-sectional area just before the tunnel inlet as compared with the cross-sectional area at the tunnel. Korean J Radiol. 2010 Nov-Dec;11(6):632-9. doi: 10.3348/kjr.2010.11.6.632. Epub 2010 Oct 29. PMID 21076589
- [Background] Chen J, Chen L, Wu L, Wang R, Liu JB, Hu B, Jiang LX. Value of superb microvascular imaging ultrasonography in the diagnosis of carpal tunnel syndrome: Compared with color Doppler and power Doppler. Medicine (Baltimore). 2017 May;96(21):e6862. doi: 10.1097/MD.0000000000006862. PMID 28538376